CLINICAL TRIAL: NCT02122913
Title: A Phase 1 Study of the Oral TRK Inhibitor Larotrectinib in Adult Patients With Solid Tumors
Brief Title: A Study to Test the Safety of the Investigational Drug Larotrectinib in Adults That May Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20288; LOXO-TRK-14001 (Other: Loxo Inc.)
Expanded Access: NCT03025360 (Approved for marketing)
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Advanced solid tumors; Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive; TRK fusion; TRKA; TRKB; TRKC; ETV6
MeSH Terms: interventions — larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Tumor patients_Dose 1 (Experimental): Adult patients with solid tumors receiving 50 mg of BAY2757556 once daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Dose 2 (Experimental): Adult patients with solid tumors receiving 100 mg of BAY2757556 once daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Dose 3 (Experimental): Adult patients with solid tumors receiving 100 mg of BAY2757556 twice daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Dose 4 (Experimental): Adult patients with solid tumors receiving 200 mg of BAY2757556 once daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Dose 5 (Experimental): Adult patients with solid tumors receiving 150 mg of BAY2757556 twice daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Dose 6 (Experimental): Adult patients with solid tumors receiving 200 mg of BAY2757556 twice daily (dose escalation cohort).
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Tumor patients_Expansion (Experimental): Adults patients with solid tumors and neurotrophic tyrosine kinase (NTRK) genes or proteins of types 1 - 3 (dose expansion cohort).
  Patients receive either the recommended or maximum tolerated dose of BAY2757556 as determined in the dose escalation part.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)

INTERVENTIONS:
Drug: Larotrectinib (Vitrakvi, BAY2757556) — BAY2757556 will be administered orally as capsule or in liquid form over continuous 28-day cycles.
  Other Names: LOXO-101

SUMMARY:
This research study is done to test the safety of the drug larotrectinib in adult cancer patients. The drug may be used to treat cancer with a change in a particular gene (NTRK1, NTRK2 or NTRK3), because it blocks the action of these genes in cancer cells. The study also investigates how the drug is absorbed and processed in the human body. This is the first study to test larotrectinib in humans with cancer, for whom no other effective therapy exists.

DETAILED DESCRIPTION:
The trial will be conducted in 2 parts: an initial dose escalation phase of larotrectinib in subjects with advanced solid tumors will be followed by an expansion phase in subjects with solid tumors having a NTRK fusion.

The objectives of the study are to determine the safety, pharmacokinetic profile, recommended dose and efficacy of orally administered larotrectinib in patients with NTRK fusions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a locally advanced or metastatic solid tumor that has progressed or was nonresponsive to available therapies, are unfit for standard chemotherapy or for which no standard or available curative therapy exists
* Proof of a malignancy harboring a NTRK fusion
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2 and a life expectancy of at least 3 months
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Patients with unstable primary central-nervous-system tumors or metastasis, exceptions possible
* Clinically significant active cardiovascular disease or history of myocardial infarction
* Active uncontrolled systemic bacterial, viral, or fungal infection
* Current treatment with a strong CYP3A4 inhibitor or inducer
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-05-04 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 25 months
Severity of adverse events | 25 months
  The severity of adverse events will be assesssed according to the NCI CTCAE version 4.03.
Maximum tolerated dose (MTD) | 25 months
Recommended dose for dose expansion | 25 months

SECONDARY OUTCOMES:
Maximum concentration of larotrectinib in plasma (Cmax) | Predose and 0.25, 0.5, 1, 2, 4, 6 and 8 hours after drug administration on Days 1 and 8 of Cycle 1
Time to maximum concentration of larotrectinib in plasma (Tmax) | Predose and 0.25, 0.5, 1, 2, 4, 6 and 8 hours after drug administration on Days 1 and 8 of Cycle 1
Half-life of larotrectinib in plasma (t1/2) | Predose and 0.25, 0.5, 1, 2, 4, 6 and 8 hours after drug administration on Days 1 and 8 of Cycle 1
Area under the concentration versus time curve of larotrectinib in plasma (AUC) | Predose and 0.25, 0.5, 1, 2, 4, 6 and 8 hours after drug administration on Days 1 and 8 of Cycle 1
Overall Response Rate (ORR) | Up to 60 months
  Assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-Oncology (RANO) as appropriate
Duration of Response (DOR) | Up to 60 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCHealth Cancer Center - Anschutz Medical Campus - University of Colorado Cancer Center, Aurora, Colorado
  - Mass General Cancer Center, Boston, Massachusetts
  - UH Seidman Cancer Center, Cleveland, Ohio
  - OHSU Hospital - Neurology, Portland, Oregon
  - Hospital of the University of Pennsylvania - Radiology, Philadelphia, Pennsylvania
  - UPMC Mercy - Oncology, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Waguespack SG, Drilon A, Lin JJ, Brose MS, McDermott R, Almubarak M, Bauman J, Casanova M, Krishnamurthy A, Kummar S, Leyvraz S, Oh DY, Park K, Sohal D, Sherman E, Norenberg R, Silvertown JD, Brega N, Hong DS, Cabanillas ME. Efficacy and safety of larotrectinib in patients with TRK fusion-positive thyroid carcinoma. Eur J Endocrinol. 2022 Apr 29;186(6):631-643. doi: 10.1530/EJE-21-1259. PMID 35333737
- [Derived] Brose MS, Westphalen CB, Pan X, Bernard-Gauthier V, Kurtinecz M, Guo H, Aris V, Brett NR, Majdi A, Subbiah V, Pennell NA, Kehl KL, Drilon A. Larotrectinib Compared With Real-World Non-Tropomyosin Receptor Kinase Inhibitor Therapies in Patients With Tropomyosin Receptor Kinase Fusion Cancer. JCO Precis Oncol. 2025 Apr;9:e2400500. doi: 10.1200/PO-24-00500. Epub 2025 Apr 23. PMID 40267388
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Kummar S, Shen L, Hong DS, McDermott R, Keedy VL, Casanova M, Demetri GD, Dowlati A, Melcon SG, Lassen UN, Leyvraz S, Liu T, Moreno V, Patel J, Patil T, Mallick AB, Sousa N, Tahara M, Ziegler DS, Norenberg R, Arvis P, Brega N, Drilon A, Tan DSW. Larotrectinib efficacy and safety in adult patients with tropomyosin receptor kinase fusion sarcomas. Cancer. 2023 Dec 1;129(23):3772-3782. doi: 10.1002/cncr.35036. Epub 2023 Sep 28. PMID 37769113
- [Derived] Bokemeyer C, Paracha N, Lassen U, Italiano A, Sullivan SD, Marian M, Brega N, Garcia-Foncillas J. Survival Outcomes of Patients With Tropomyosin Receptor Kinase Fusion-Positive Cancer Receiving Larotrectinib Versus Standard of Care: A Matching-Adjusted Indirect Comparison Using Real-World Data. JCO Precis Oncol. 2023 Jan;7:e2200436. doi: 10.1200/PO.22.00436. PMID 36689698
- [Derived] Rudzinski ER, Drilon A, Moore A, Spinosa S, Willi M, Laetsch TW. Testing methods to diagnose TRK fusion cancer - a plain language summary and patient perspective. Future Oncol. 2022 Dec;18(38):4141-4151. doi: 10.2217/fon-2022-0863. Epub 2023 Jan 6. PMID 36606522
- [Derived] Le X, Baik C, Bauman J, Gilbert J, Brose MS, Grilley-Olson JE, Patil T, McDermott R, Raez LE, Johnson JM, Shen L, Tahara M, Ho AL, Norenberg R, Dima L, Brega N, Drilon A, Hong DS. Larotrectinib Treatment for Patients With TRK Fusion-Positive Salivary Gland Cancers. Oncologist. 2022 May 10;29(6):e779-88. doi: 10.1093/oncolo/oyac080. Online ahead of print. PMID 35536733
- [Derived] Drilon A, Tan DSW, Lassen UN, Leyvraz S, Liu Y, Patel JD, Rosen L, Solomon B, Norenberg R, Dima L, Brega N, Shen L, Moreno V, Kummar S, Lin JJ. Efficacy and Safety of Larotrectinib in Patients With Tropomyosin Receptor Kinase Fusion-Positive Lung Cancers. JCO Precis Oncol. 2022 Jan;6:e2100418. doi: 10.1200/PO.21.00418. PMID 35085007
- [Derived] Bebb DG, Banerji S, Blais N, Desmeules P, Gill S, Grin A, Feilotter H, Hansen AR, Hyrcza M, Krzyzanowska M, Melosky B, Noujaim J, Purgina B, Ruether D, Simmons CE, Soulieres D, Torlakovic EE, Tsao MS. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Adults. Curr Oncol. 2021 Jan 15;28(1):523-548. doi: 10.3390/curroncol28010053. PMID 33467570
- [Derived] Perreault S, Chami R, Deyell RJ, El Demellawy D, Ellezam B, Jabado N, Morgenstern DA, Narendran A, Sorensen PHB, Wasserman JD, Yip S. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Pediatric Patients. Curr Oncol. 2021 Jan 9;28(1):346-366. doi: 10.3390/curroncol28010038. PMID 33435412
- [Derived] Hong DS, DuBois SG, Kummar S, Farago AF, Albert CM, Rohrberg KS, van Tilburg CM, Nagasubramanian R, Berlin JD, Federman N, Mascarenhas L, Geoerger B, Dowlati A, Pappo AS, Bielack S, Doz F, McDermott R, Patel JD, Schilder RJ, Tahara M, Pfister SM, Witt O, Ladanyi M, Rudzinski ER, Nanda S, Childs BH, Laetsch TW, Hyman DM, Drilon A. Larotrectinib in patients with TRK fusion-positive solid tumours: a pooled analysis of three phase 1/2 clinical trials. Lancet Oncol. 2020 Apr;21(4):531-540. doi: 10.1016/S1470-2045(19)30856-3. Epub 2020 Feb 24. PMID 32105622
- [Derived] Hong DS, Bauer TM, Lee JJ, Dowlati A, Brose MS, Farago AF, Taylor M, Shaw AT, Montez S, Meric-Bernstam F, Smith S, Tuch BB, Ebata K, Cruickshank S, Cox MC, Burris HA 3rd, Doebele RC. Larotrectinib in adult patients with solid tumours: a multi-centre, open-label, phase I dose-escalation study. Ann Oncol. 2019 Feb 1;30(2):325-331. doi: 10.1093/annonc/mdy539. PMID 30624546
- [Derived] Drilon A, Laetsch TW, Kummar S, DuBois SG, Lassen UN, Demetri GD, Nathenson M, Doebele RC, Farago AF, Pappo AS, Turpin B, Dowlati A, Brose MS, Mascarenhas L, Federman N, Berlin J, El-Deiry WS, Baik C, Deeken J, Boni V, Nagasubramanian R, Taylor M, Rudzinski ER, Meric-Bernstam F, Sohal DPS, Ma PC, Raez LE, Hechtman JF, Benayed R, Ladanyi M, Tuch BB, Ebata K, Cruickshank S, Ku NC, Cox MC, Hawkins DS, Hong DS, Hyman DM. Efficacy of Larotrectinib in TRK Fusion-Positive Cancers in Adults and Children. N Engl J Med. 2018 Feb 22;378(8):731-739. doi: 10.1056/NEJMoa1714448. PMID 29466156
- [Derived] Doebele RC, Davis LE, Vaishnavi A, Le AT, Estrada-Bernal A, Keysar S, Jimeno A, Varella-Garcia M, Aisner DL, Li Y, Stephens PJ, Morosini D, Tuch BB, Fernandes M, Nanda N, Low JA. An Oncogenic NTRK Fusion in a Patient with Soft-Tissue Sarcoma with Response to the Tropomyosin-Related Kinase Inhibitor LOXO-101. Cancer Discov. 2015 Oct;5(10):1049-57. doi: 10.1158/2159-8290.CD-15-0443. Epub 2015 Jul 27. PMID 26216294
- See also: A plain language summary of two trials for larotrectinib in people with TRK fusion-positive lung cancer to learn how well the drug works and how safe it is — https://pubmed.ncbi.nlm.nih.gov/40539316/
- See also: Testing methods to diagnose TRK fusion cancer - a plain language summary and patient perspective — https://pubmed.ncbi.nlm.nih.gov/36606522/